CLINICAL TRIAL: NCT06704477
Title: Dietary Protein Preferences of Adolescent Athletes
Status: Completed | Type: Observational
Sponsor: PepsiCo Global R&D (Industry)
Responsible Party: Sponsor
Other Study IDs: PEP-2310
Record Dates: First submitted 2024-11-22; First posted 2024-11-26 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2025-01

CONDITIONS: Diet Habit
Keywords: protein; animal protein; plant protein; preference
MeSH Terms: conditions — Feeding Behavior | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Survey — Eight questions about protein intake

SUMMARY:
This is a survey study to gauge the interest of young athletes ages 12-19 in plant-based protein products. The teen competitive athlete is a core target for the Gatorade brand and, as such, understanding their preferences and what drives their choices is vital for the brand's continued growth.

ELIGIBILITY:
Inclusion Criteria:

* Male and female student-athletes between the ages of 12-19 years
* Athlete must currently participate in a sport at the middle/high school level
* Athlete must be able to speak, write, and read English
* Athlete must own a smartphone with access to internet and text message service (to complete survey)
* Athlete (and parent/guardian, if under 18 years of age) must understand the study procedures and be willing to sign the informed consent form providing consent/assent to participate in the stud

Exclusion Criteria:

• Athlete must not be employed by, or have a parent, guardian, or other immediate family member employed by a company that manufactures any products that compete with any Gatorade product

Ages: 12 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Student athletes
Sampling Method: Non-Probability Sample
Enrollment: 161 (Actual)
Dates: Start 2024-02-22 (Actual); Primary Completion 2024-10-25 (Actual); Study Completion 2024-10-25 (Actual)

PRIMARY OUTCOMES:
Most preferred protein type in adolescent athletes (i.e. animal vs. plant protein) | Each participant has three (3) weeks to open/complete the survey from time of receipt. Participants will be instructed to complete the survey in one sitting during a time and in an environment in which they can fully devote their attention and focus.
  Part of a 10 minute multiple choice survey

SECONDARY OUTCOMES:
Reported reason(s) for protein preference | Each participant has three (3) weeks to open/complete the survey from time of receipt. Participants will be instructed to complete the survey in one sitting during a time and in an environment in which they can fully devote their attention and focus.
  Part of a 10 minute multiple choice survey
% of athletes who consume protein supplements | Each participant has three (3) weeks to open/complete the survey from time of receipt. Participants will be instructed to complete the survey in one sitting during a time and in an environment in which they can fully devote their attention and focus.
  Part of a 10 minute multiple choice survey
Specific type(s) of protein supplement source(s) consumed (soy, pea, whey, casein, etc.) | Each participant has three (3) weeks to open/complete the survey from time of receipt. Participants will be instructed to complete the survey in one sitting during a time and in an environment in which they can fully devote their attention and focus.
  Part of a 10 minute multiple choice survey
Breakdown and differences by gender | Each participant has three (3) weeks to open/complete the survey from time of receipt. Participants will be instructed to complete the survey in one sitting during a time and in an environment in which they can fully devote their attention and focus.
  Part of a 10 minute multiple choice survey
Timing(s) of daily protein consumption | Each participant has three (3) weeks to open/complete the survey from time of receipt. Participants will be instructed to complete the survey in one sitting during a time and in an environment in which they can fully devote their attention and focus.
  Part of a 10 minute multiple choice survey
Most valued protein supplement attribute(s) (taste, protein, amount, source, etc.) | Each participant has three (3) weeks to open/complete the survey from time of receipt. Participants will be instructed to complete the survey in one sitting during a time and in an environment in which they can fully devote their attention and focus.
  Part of a 10 minute multiple choice survey

CONTACTS AND LOCATIONS:
Overall Officials: Khalil Lee, PhD, Principal Investigator — PepsiCo, Inc. Sports Science
Locations (1):
- IMG Academy, Bradenton, Florida, United States

IPD SHARING:
Plan to Share IPD: No